CLINICAL TRIAL: NCT04031261
Title: National Validation and Sensitivity to Change of a Scale to Measure Quality of Life in Patients With Severe Asthma
Brief Title: National Validation and Sensitivity to Change of the SAQ
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: 18/P/089
Record Dates: First submitted 2019-06-28; First posted 2019-07-24 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2019-06

CONDITIONS: Asthma; Severe Asthma
Keywords: Quality of Life; Patient Reported Outcomes
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- National Validation: All patients must have a diagnosis of severe asthma, be taking high dose inhaled corticosteroids (GINA step 4 & 5), and be aged 16 years or over.
- Sensitivity to Change: Patients commencing a biologic treatment for their severe asthma (GINA step 4 & 5), as per National Institute for Health and Care Excellence (NICE) guidelines.

SUMMARY:
DESIGN A multi-centre mixed methods study of a new asthma specific quality of life questionnaire including limited clinic data.

AIMS To collect further quantitative data to validate a new asthma quality of life scale, the Severe Asthma Questionnaire (SAQ).

To determine the Minimum Clinically Important Difference (MCID) of the SAQ

OUTCOME MEASURES

Questionnaires:

1. The Severe Asthma Questionnaire (SAQ)
2. The Mini Asthma Quality of Life Questionnaire (MiniAQLQ)
3. The EQ-5D-5L
4. The Asthma Control Test (ACT)/ Asthma Control Questionnaire (ACQ)
5. Global Rating of Change Questionnaire (GRCQ)

   Clinical data comprises:
6. Spirometry
7. BMI
8. Asthma severity
9. Health care utilisation: ED attendance in the last 12 months, Hospital admissions in the last 12 months;
10. Number of exacerbations in the last 12 months requiring OCS Prednisolone dose mg/day (if oral steroid dependent).

POPULATION All patients aged 16 years or over, who have attended one of three participating UK specialist asthma centres for the validation study and with data also collected from Derriford Hospital's Chest Clinic (DHCC) for use in determining Minimum clinically Important difference.

ELIGIBILITY Over 16 years of age Diagnosis of Severe Asthma

DURATION 18 months

ELIGIBILITY:
Part 1: National Validation

Inclusion Criteria:

* All patients must have a diagnosis of severe asthma, be taking high dose inhaled corticosteroids (GINA step 4 & 5), and be aged 16 years or over.

Exclusion Criteria:

* Patients that are unwilling to participate will be excluded from the study.
* In the opinion of the physician responsible for the care of the patient, the patient has a condition, other than asthma, which is significantly contributing to their respiratory symptoms, e.g. lung cancer, heart failure or severe Chronic Obstructive Pulmonary Disease (COPD).
* The SAQ is currently only translated into British English. Therefore, if the participant is unable to read in English, they will be unable to participate.

Part 2: Sensitivity to change

Inclusion Criteria

* Patients commencing a biologic treatment for their severe asthma (GINA step 4 & 5), as per NICE guidelines.

Exclusion Criteria

* Patients will be excluded from the study if they are unwilling to participate
* In the opinion of the physician responsible for the care of the patient, the patient has a condition, other than asthma which is significantly contributing to their respiratory symptoms, e.g. lung cancer, heart failure or severe COPD.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients must have a diagnosis of severe asthma, be taking high dose inhaled corticosteroids (GINA step 4 & 5), and be aged 16 years or over.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Severe Asthma Questionnaire (SAQ) score | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment (enrollment period of 6 months)
  The new questionnaire will provide a combined assessment of disease and its treatment on the quality of life of patients with severe asthma. The scale is based on existing Health Related Quality of Life (HRQoL) scales but modified for the severe population and provides assessments of the effect of asthma symptoms and the effect of asthma medicines. The SAQ was produced from detailed qualitative research. The questionnaire has 16 items, scored on a 1-7 scale (a higher score indicating better quality of life). The mean score of these 16 questions is calculated to produce an overall score.
  An additional 3 items are included to asses overall HRQoL, and HRQoL during different months of the year. These three questions are scored on a 100 point scale with a higher score indicating better HRQoL.
Change in Severe Asthma Questionnaire (SAQ) score | Part 2: Sensitivity to change: Collected at 0 (baseline) 4, 8, 12 & 16 weeks, (enrollment period of 10 months)
  The Severe Asthma Questionnaire (SAQ) will be collected at 5 time points and matched with the Global Rating of Change questionnaire at these time points to determine the SAQ's Minimum Clinically Important Difference (MCID).
  The questionnaire has 16 items, scored on a 1-7 scale (a higher score indicating better quality of life). The mean score of these 16 questions is calculated to produce an overall score.
  An additional 3 items are included to asses overall HRQoL, and HRQoL during different months of the year. These three questions are scored on a 100 point scale with a higher score indicating better HRQoL.

SECONDARY OUTCOMES:
The Mini Asthma Quality of Life Questionnaire (MiniAQLQ) | Part 1: National Validation & Part 2: Sensitivity to change - Collected at 0 (baseline) weeks, within two weeks after enrollment (enrollment period of 6 or 10 months respectively)
  This 15-item scale is commonly used as the quality of life scale in asthma studies. It consists of 15 questions which are scored on on a 1-7 scale, with a higher score indicating better health related quality of life. Whilst the MiniAQLQ can be scored as four separate domains (Symptoms, Activity Limitations, Emotional Functional and Environmental Stimuli), these will not be used. Instead the mean score of the 15 questions will be used as the MiniAQLQ score.
  For the purpose of validation, we wish to show that this scale correlates with the burden of symptoms but not, or with a much lower correlation, with the burden of treatment.
Asthma Control Test (ACT) | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment (enrollment period of 6 months), Part 2: Sensitivity to change - Collected at 0 (baseline) 4, 8, 12 & 16 weeks
  Note: Recruiting sites are able to chose which Asthma Control Patient Reported Outcome (PRO) to contribute data for, (The ACT or the ACQ).
  The Asthma Control Test (ACT) is a 5-item scale is commonly used as a measure of asthma control in asthma studies. It is scored on a scale of 1-5 with a higher score indicating better asthma control. For the purpose of validation, we wish to show that this scale correlates with the burden of symptoms but not, or with a much lower correlation, with the burden of treatment.
Asthma Control Questionnaire (ACQ) | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline) 4, 8, 12 & 16 weeks
  The Asthma Control Questionnaire (ACQ) contains 7 items and takes into consideration FEV1% predicted and daily use of rescue bronchodilator. Patients respond to 7 items concerning their symptom severity on a 0-6 scale (0 = no impairment, 6 = maximum impairment). The mean of the 7-items will be used as the score of the ACQ.
EQ-5D-5L | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment (enrollment period of 6 months) , Part 2: Sensitivity to change - Collected at 0 (baseline) & 16 weeks within 2 weeks of enrollment
  This is a 5-item scale scored from 1-5 with a higher score indicating worse health. For the purposes of this study, the mean score of the five items will be used as the score for the EQ5D. In addition to the 5 items, the EQ-5D-5L also includes a category rating scale to rate their quality of life on the day of completion. This is scored from 0-100 with a higher score indicating better health.
  This scale is commonly used in clinical trials to determine improvement in patients' perceived quality of life.
  The correlations between EQ-5D-5L scores and SAQ scores will be explored.
Change in Global Rating of Change Questionnaire (GRCQ) | Part 2: Sensitivity to change - Collected at 4, 8, 12 & 16 weeks within 2 weeks of enrollment (enrollment period of 10 months)
  This scale will be used by participants to indicate how much better they feel since commencing a biologic treatment for asthma. The 11-point scale ranges from -5 (a great deal worse) to 5 (A great deal better).

OTHER OUTCOMES:
Forced Expiatory Volume in One Second (FEV1) | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline) & 16 weeks
Percentage of predicted FEV1 (FEV1%) | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline) & 16 weeks
Body Mass Index (BMI) | Part 1: National Validation & Part 2: Sensitivity to change - Collected at 0 (baseline) weeks, within two weeks after enrollment (enrollment period of 6 or 10 months respectively)
Maintenance Oral Corticosteroid dose (mg/day) | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline) 4, 8, 12 & 16 weeks
  If a participant is prescribed a daily dose of Oral Corticosteroids (OCS), this and the dose will be recorded.
  Any change to this dose will be recorded for the duration of the data collection period of part 2 of this study.
Number of exacerbation in the last 12 months requiring OCS | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline). Additional exacerbation since baseline recorded at 4, 8, 12 & 16 weeks
Number of Emergency Department attendances in the last 12 months | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline). Additional ED visits 0 since baseline recorded at 4, 8, 12 & 16 weeks
Number Hospital admissions in the last 12 months | Part 1: National Validation - Only cross-sectional data recorded within 2 weeks after enrollment, Part 2: Sensitivity to change - Collected at 0 (baseline). Additional Hospital admissions since baseline recorded at 4, 8, 12 & 16 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Devon & Exeter Hospital, Exeter
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital - Manchester, Manchester
  - University Hopsitals Plymouth NHS Trust, Plymouth

DOCUMENTS (1):
  • Study Protocol (2019-05-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT04031261/Prot_000.pdf